CLINICAL TRIAL: NCT01074658
Title: CoreValve Advance International Post Market Study: Evaluation of the Medtronic CoreValve System in a "Real-World" Patient Population.
Brief Title: CoreValve Advance International Post Market Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: Advance
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Severe Aortic Stenosis
Keywords: Advance; Medtronic CoreValve System; International; Interventional; Post Market Study
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- severe aortic valve stenosis: elderly patients with severe aortic valve stenosis requiring treatment
  Interventions: Device: Medtronic CoreValve System

INTERVENTIONS:
Device: Medtronic CoreValve System — Transcatheter Aortic Valve Implantation of the Medtronic CoreValve System

SUMMARY:
The CoreValve Advance study is intended to evaluate the clinical utility of the Medtronic CoreValve System in a "Real-World" patient population.

DETAILED DESCRIPTION:
The CoreValve Advance study is intended to evaluate the clinical utility of the Medtronic CoreValve System for percutaneous aortic valve implantation in a "Real-World" patient population with severe aortic valve stenosis. Data collected in this study will provide additional information on the understanding of the safety and device performance and how to best treat elderly patients with severe aortic valve stenosis. In addition, health economic data will be collected to understand the improvement of quality of life and the cost effectiveness of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe aortic valve stenosis requiring treatment
* Patient is an acceptable candidate for elective treatment with the Medtronic CoreValve System and in conformity with the local regulatory and medico economical context
* Patient is above the minimum age as required by local regulations to be participating in a clinical study
* The patient or legal representative has been informed of the nature of the study and has consented to participate, and has authorized the collection and release of his/her medical information by signing a consent form ("Patient Informed Consent Form")

Exclusion Criteria:

* Currently participating in another trial
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with severe aortic valve stenosis requiring treatment, who are selected to be treated electively with the Medtronic CoreValve System
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Linke, Prof Dr med, Principal Investigator — Universitat Leipzig Herzzentrum
Locations (44):
- Belgium (3):
  - ZNA Antwerpen Middelheim, Antwerp
  - Antwerpen UZA, Antwerp
  - CHU Sart Tillman, Liège
- Angiografia de Occidente, Cali, Colombia
- Rigshospitalet, Copenhagen, Denmark
- France (6):
  - Hopital Henri Mondor, Créteil
  - Hopital Cardiologique, Lille
  - Hopital Louis Pradel, Lyon
  - Institut Hospitalier Jacques Cartier, Massy
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Clinique Pasteur, Toulouse
- Germany (7):
  - Universitätsklinikum Aachen, Aachen
  - Bernau Herzzentrum Brandenburg, Bernau B. Berlin
  - CardioVascular Center Frankfurt, Frankfurt
  - Asklepios Klinik St. Georg Hamburg, Hamburg
  - Universitat Leipzig Herzzentrum, Leipzig
  - Deutsches Herzzentrum Munchen, München
  - Helios Herzzentrum Siegburg Gmbh, Siegburg
- Onassis cardiac surgery center, Athens, Greece
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Tel Aviv
  - Ichilov Medical Center, Tel Aviv
- Italy (8):
  - Azienda Ospedaliere Spedali Civili di Brescia, Brescia
  - Policlinico Vittorio Emanuele, P.O. Ferrarotto, Catania
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Civile, Legnano
  - Ospedale Niguarda Ca'Granda, Milan
  - Fondazione Centro San Raffaele, Milan
  - Istituto Clinico S.Ambrogio, Milan
  - Istituto Clinico Humanitas, Rozzano
- Netherlands (4):
  - AMC Ziekenhuis, Amsterdam
  - Amphia Breda, Breda
  - Catharina Hospital, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
- Portugal (2):
  - Hospital de Santa Cruz, Lisbon
  - Centro Hospitalar de Vila Nova de Gaia, Porto
- Switzerland (2):
  - Universtiy Hospital Isel Bern, Bern
  - Universitätsspital Zürich, Zurich
- United Kingdom (6):
  - Brighton and Sussex Hospital, Brighton
  - Leeds General Infirmary, Leeds
  - Leicester Hospital, Leicester
  - St. George's Hospital, London
  - The Heart Hospital, London
  - Newcross Hospital Wolverhampton, Wolverhampton

REFERENCES:
- [Derived] Gerckens U, Tamburino C, Bleiziffer S, Bosmans J, Wenaweser P, Brecker S, Guo J, Linke A. Final 5-year clinical and echocardiographic results for treatment of severe aortic stenosis with a self-expanding bioprosthesis from the ADVANCE Study. Eur Heart J. 2017 Sep 21;38(36):2729-2738. doi: 10.1093/eurheartj/ehx295. PMID 28633375
- [Derived] Bleiziffer S, Bosmans J, Brecker S, Gerckens U, Wenaweser P, Tamburino C, Linke A; ADVANCE Study Investigators. Insights on mid-term TAVR performance: 3-year clinical and echocardiographic results from the CoreValve ADVANCE study. Clin Res Cardiol. 2017 Oct;106(10):784-795. doi: 10.1007/s00392-017-1120-3. Epub 2017 May 8. PMID 28484830
- [Derived] Brecker SJ, Bleiziffer S, Bosmans J, Gerckens U, Tamburino C, Wenaweser P, Linke A; ADVANCE Study Investigators. Impact of Anesthesia Type on Outcomes of Transcatheter Aortic Valve Implantation (from the Multicenter ADVANCE Study). Am J Cardiol. 2016 Apr 15;117(8):1332-8. doi: 10.1016/j.amjcard.2016.01.027. Epub 2016 Jan 28. PMID 26892451
- [Derived] Barbanti M, Schiltgen M, Verdoliva S, Bosmans J, Bleiziffer S, Gerckens U, Wenaweser P, Brecker S, Gulino S, Tamburino C, Linke A; ADVANCE Study Investigators. Three-Year Outcomes of Transcatheter Aortic Valve Implantation in Patients With Varying Levels of Surgical Risk (from the CoreValve ADVANCE Study). Am J Cardiol. 2016 Mar 1;117(5):820-7. doi: 10.1016/j.amjcard.2015.11.066. Epub 2015 Dec 13. PMID 26762727
- [Derived] Bosmans J, Bleiziffer S, Gerckens U, Wenaweser P, Brecker S, Tamburino C, Linke A; ADVANCE Study Investigators. The Incidence and Predictors of Early- and Mid-Term Clinically Relevant Neurological Events After Transcatheter Aortic Valve Replacement in Real-World Patients. J Am Coll Cardiol. 2015 Jul 21;66(3):209-217. doi: 10.1016/j.jacc.2015.05.025. PMID 26184612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start Recruitment March 2010 > End Recruitment July 2011
Groups:
- Medtronic CoreValve System: Transcatheter Aortic Valve Implantation (TAVI) with the Medtronic CoreValve System.
Period: Overall Study
Arm/Group | Medtronic CoreValve System
Started | 1015
Attempted Implant | 996
Completed | 996
Not Completed | 19
Not completed — No implant attempted | 19

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic CoreValve System
Number analyzed (Participants) | 1015
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 514
  Male | 501

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac & Cerebrovascular Events (MACCE)
Description: MACCE is defined as a composite of:
  * All cause mortality
  * Myocardial Infarction (Q-wave and non-Q-wave)
  * Emergent cardiac surgery or percutaneous re-intervention
  * Stroke
  The Kaplan-Meier survival analysis was used to derive the freedom from MACCE at 30 days.
Time Frame: 30 days
Population: All attempted population.
Measure: Number; unit: Freedom from MACCE (%) @30days
Arm/Group | Medtronic CoreValve System
Number analyzed (Participants) | 996
Freedom from MACCE (%) @30days | 92

2. Secondary Outcome: Percentage of Participants With Device Success
Description: Device Success is defined as a composite of:
  * Successful device delivery;
  * Stable device placement;
  * Intact retrieval of delivery catheter;
  * Successful device function as assessed immediately post-procedure by angiography including non-compromised flow in coronary arteries (without obstruction) device position (no migration) and a mean gradient as determined invasively of <15mmHg and ≤ 2 aortic regurgitation
Time Frame: up to 24 hours
Population: All attempted population in which the separate variables related to device success (see outcome measure description) were analyzable.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve System
Number analyzed (Participants) | 578
percentage of participants | 79.4

3. Secondary Outcome: Percentage of Participants With Procedural Success
Description: Procedural success, defined as device success with absence of in-hospital MACCE
Time Frame: up to 30 days
Population: All attempted population in which the separate variables related to procedural success (see outcome measure description) were analyzable.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve System
Number analyzed (Participants) | 613
percentage of participants | 71.1

ADVERSE EVENTS:
Time Frame: 30 days post procedure
Arm/Group | Medtronic CoreValve System
Serious Adverse Events (participants affected / at risk) | 541/996
Other Adverse Events (participants affected / at risk) | 541/996
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic CoreValve System (N=996)
Cardiac tamponade (Cardiac disorders) | 3 (3)
Vessel dissection (Injury, poisoning and procedural complications) | 4 (4)
Access site complication (Injury, poisoning and procedural complications) | 6 (6)
Access vessel dissection (Injury, poisoning and procedural complications) | 21 (21)
Access vessel perforation (Injury, poisoning and procedural complications) | 15 (15)
Acute vessel occlusion (Injury, poisoning and procedural complications) | 7 (7)
Hemorrhage requiring transfusion (Injury, poisoning and procedural complications) | 9 (9)
Bradycardia (Cardiac disorders) | 4 (4)
Reposition with snare (Injury, poisoning and procedural complications) | 2 (2)
Valve in valve (Injury, poisoning and procedural complications) | 15 (15)
Valve retrieval (Injury, poisoning and procedural complications) | 4 (4)
Valve dislocation into LVOT (Injury, poisoning and procedural complications) | 1 (1)
Valve dislocation into annular aorta (Injury, poisoning and procedural complications) | 6 (6)
Ventricular rupture (Injury, poisoning and procedural complications) | 3 (3)
Hemodynamic instability requiring Heart/Lung machine (Vascular disorders) | 2 (2)
Resuscitation (Surgical and medical procedures) | 9 (9)
Ventricular fibrillation (Cardiac disorders) | 6 (6)
Failure of closure device requiring surgery (Surgical and medical procedures) | 11 (11)
Arrhythmia (Cardiac disorders) | 18 (18)
Other Procedural Complication (Injury, poisoning and procedural complications) | 23 (25)
Death (General disorders) | 45 (45)
Stroke/TIA (Nervous system disorders) | 30 (30)
Myocardial Infarction (Cardiac disorders) | 110 (110) — Myocardial infarction was defined according to the definition proposed by the The Joint ESC/ACC/AHA/WHF Task Force and Academic Research Consortium.(Thygesen K, Alpert JS, White HD. Circulation. 2007;116:2634-2653)
Renal Failure (Renal and urinary disorders) | 35 (36)
Structural Valve Deterioration (Cardiac disorders) | 1 (1)
Nonstructural Valve Dysfunction (Cardiac disorders) | 7 (7)
Bleeding Event (Vascular disorders) | 87 (91) — Any episode of major internal or external bleeding that causes death, hospitalization, or permanent injury (i.e. vision loss) or necessitates transfusion.
Permanent Pacemaker Implantation (Surgical and medical procedures) | 209 (209)
Other Serious Adverse Event (General disorders) | 213 (286)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic CoreValve System (N=996)
AE related to Device (General disorders) | 84 (101)
AE related to Index procedure (General disorders) | 535 (883)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI will provide results to sponsor for review and approval at least 60 days prior to submittal for publication or presentation. Review will be limited to determination whether Confidential Information is disclosed and not to censor or interfere with presentation or conclusions beyond the extent necessary to protect Confidential Information, to allow the sponsor to protect its rights in patentable or copyrightable material, and to check for technical correctness of sponsor information.